CLINICAL TRIAL: NCT07251972
Title: Comparison of Two Methods of Immunoprophylaxis Against RSV in Term Newborns in a Level 3 Maternity Unit During Winter 2025-2026
Brief Title: Comparison of Two Methods of Immunoprophylaxis Against RSV in Term Newborns
Acronym: Abrystus
Status: Active, not recruiting | Type: Observational
Sponsor: Jean-Michel HASCOET (Other)
Responsible Party: Sponsor-Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2025PI033
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Bronchiolitis
Keywords: immunoprophylaxis RSV
MeSH Terms: conditions — Bronchiolitis | interventions — Antibodies, Monoclonal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: to compare vaccine and monoclonal antibody — collect the details at birth of chosen immunoprophylaxis and collect if later there will be any hospitalisation for bronchiolitis or consultation emergencies

SUMMARY:
Bronchiolitis is a lower respiratory tract infection, extremely common in pediatrics, and potentially serious. Bronchiolitis affects nearly 30% of infants under 2 years old each year, representing approximately 480,000 cases annually worldwide. Each year, 2 to 3% of infants under 1 year old are hospitalized for bronchiolitis. The virus primarily found worldwide and in France is RSV. Given the scale, frequency, and potential severity of the illness, several immunoprophylaxis methods have been developed.

Currently, there are two methods: the ABRYSVO vaccine, administered to pregnant women during the last month of pregnancy for immunization via the placenta through the transplacental passage of anti-RSV-A and RSV-B antibodies; or neonatal immunoprophylaxis with BEYFORTUS, which involves an intramuscular injection of the monoclonal antibody nirvesimab directly into the newborn immediately before discharge from the maternity ward during the epidemic period.

Currently, no superiority or difference has been described for either immunoprophylaxis method.

ELIGIBILITY:
Inclusion Criteria:

* all term born neonates

Exclusion Criteria:

* postnatal transfert
* born at home or in birthing center

Ages: 4 Days to 8 Months | Sex: All
Age Groups: Child
Study Population: term born neonate
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Bronchiolitis incidence | 8 months
  Number of emergency room visits for bronchiolitis

CONTACTS AND LOCATIONS:
Locations (1):
- Chru Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No